CLINICAL TRIAL: NCT00470457
Title: A Randomized Study to Evaluate a Novel Method of Specific Allergen Immunotherapy in Grass and/or Tree Pollen Allergic Subjects by Intralymphatic Allergen Administration
Brief Title: A Randomized Study to Evaluate a Novel Method of Specific Allergen Immunotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: AlleCure (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-GTP-001
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Rhinoconjunctivitis Due to Grass Pollen Allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Allergen specific immunotherapy

SUMMARY:
Allergen specific immunotherapy (SIT) is the only causative treatment of IgE-mediated allergies. The disadvantages of SIT, however, are the requirement of numerous allergen administrations over three to five years, and that the treatment itself causes frequent allergic reactions. We aim at enhancing grass pollen SIT in hay fever patients by injecting the allergen directly into subcutaneous lymph nodes. In a monocentric randomized trial safety and efficacy of intralymphatic immunotherapy (ILIT) with 3 low dose grass pollen extract injections over 2 months are compared to subcutaneous immunotherapy (SCIT) using 54 injections over 3 years.

* Trial with immunodulatory product / biological

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* History of allergic rhino-conjunctivitis in spring and summer
* Age 18 years to 65 years
* Positive skin prick test to grass pollen

Exclusion criteria:

* Blood donation within previous 30 days
* Surgery within the previous 30 days
* Use of investigational drugs within previous 90 days
* Pregnancy or nursing
* Mastocytosis
* Significant cardiovascular disease
* Hypertension
* Active infectious disease
* Significant hepatic disease
* Significant renal disease
* Significant hematological disorder
* Significant pulmonary disease
* Moderate or severe asthma
* Autoimmune disease
* History of malignancy.
* Contraindicated medications were immunosuppressive agents, beta-blockers, ACE-inhibitors, and tricyclic antidepressants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2001-06; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Safety efficacy and toxicity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Clinic for Dermatology University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265